CLINICAL TRIAL: NCT05500560
Title: Effect of COVID-19 on Endothelial Function
Status: Completed | Type: Observational
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Athanasios Moulias, Principal Investigator, University Hospital of Patras
Other Study IDs: 16/02-02-2022
Record Dates: First submitted 2022-07-30; First posted 2022-08-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; Endothelial Dysfunction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Patients admitted to our hospital due to COVID-19
- Controls: Healthy volunteers matched for age, sex and cardiovascular risk factors.

SUMMARY:
COVID-19 disease (coronavirus disease 2019) primarily affects the respiratory system, using the angiotensin-converting enzyme 2 receptor. However, there is increasing evidence that COVID-19 can also affect the heart (myocardial injury, myocarditis, arrhythmias) and the vascular system, effects that may worsen the clinical outcome of patients.

The aim of this study is to assess the effect of COVID-19 on the patients' endothelial function, during the acute phase of the disease (inpatient), shortly after recovery (2 months) and in the mid-term (6 months). Evaluation of endothelial function will be performed non-invasively by the method of Peripheral Arterial Tonometry (PAT) using the EndoPAT2000 system (Itamar Medical, Israel).

This is a prospective, case-controlled, single-center clinical observational study.

The study will include adult patients who developed COVID-19 disease for whom admission for hospitalization was required, while the control group will consist of healthy volunteers matched for age, gender and cardiovascular risk factors.

Patients enrolled in the study will undergo the following visits:

* Visit 1: Hospitalization
* Visit 2: 2 months after discharge
* Visit 3: 6 months after discharge
* Visit 4: 1 year after discharge Patients will be subjected to measurement of the reactive hyperemia index with the EndoPAT2000 system in Visits 1, 2 and 3.

The aim of the study is to compare the endothelial function between the two groups (COVID-19 vs. Controls).

DETAILED DESCRIPTION:
1. Introduction COVID-19 disease (coronavirus disease 2019) primarily affects the respiratory system, using the angiotensin-converting enzyme 2 receptor. However, there is increasing evidence that COVID-19 can also affect the heart (myocardial injury, myocarditis, arrhythmias) and the vascular system, effects that may worsen the clinical outcome of patients.

   Regarding COVID-19, there is increasing evidence of endothelial dysfunction, both directly due to direct infection of the vascular endothelium by the SARS-COV-2 virus (endothelitis), and indirectly due to the systemic inflammatory response and cascade of cytokines.

   In the context of this study, the evaluation of endothelial function will be performed non-invasively by the method of Peripheral Arterial Tonometry (PAT) using the EndoPAT2000 system (Itamar Medical, Israel). The EndoPAT system quantifies the endothelium-dependent pulsatile arterial volume changes. During the examination, plethysmography biosensors are placed in the right and left patient's index fingers. Subsequently, arterial tone is measured in three phases:

   A. at rest (baseline) B. during ischemia caused by a cuff inflated in one of the two arms at a level above that of systolic blood pressure for a period of 5 minutes C. during the phase of reactive hyperemia after the lifting of the arterial blockade by deflating the cuff The arterial tone signals detected in the above phases of the examination by the plethysmography biosensors are converted into digital signals for each upper limb and the EndoPAT2000 system software finally calculates the hyperemic vascular response (Ln Reactive Hyperemia Index-LnRHI). Endothelial dysfunction is defined as LnRHI≤0.51.
2. Aim of the study The aim of this study is to assess the effect of COVID-19 on the patients' endothelial function, during the acute phase of the disease (inpatient), shortly after recovery (2 months) and in the mid-term (6 months).
3. Methods This is a prospective, case-controlled, single-center clinical observational study.

The study will include adult patients who developed COVID-19 disease for whom admission for hospitalization was required, while the control group will consist of healthy volunteers matched for age, gender and cardiovascular risk factors.

Based on the limited existing data, patients in the COVID group are expected to have an average LnRHI of 0.58 (SD 0.25) at 2 months after discharge versus an average LnRHI of 0.79 in the control group. By selecting α=0.05, power=90% and enrollment ratio=1, the inclusion of 30 patients in each group is required to detect the above difference (60 in total).

Patients enrolled in the study will undergo the following visits:

* Visit 1: Hospitalization
* Visit 2: 2 months after discharge
* Visit 3: 6 months after discharge
* Visit 4: 1 year after discharge Patients will be subjected to measurement of the reactive hyperemia index with the EndoPAT2000 system in Visits 1, 2 and 3.

For all participants, the following will also be recorded:

* Demographics, cardiovascular risk factors, past medical history, chronic medical treatment
* Body weight, body mass index (BMI), systolic and diastolic blood pressure, resting heart rate
* Laboratory testing: Ht, Hgb, PLT, WBC, Ur, Cr, K, Na, SGOT, SGPT, UA, total cholesterol, LDL cholesterol, small dense LDL cholesterol, HDL cholesterol, triglycerides, non-HDL cholesterol, fasting glucose, HbA1c, insulin, hsCRP, thyroid function check (TSH, T3, fT4), hs Troponin I
* ECG
* Thansthoracic ultrasound study (LVEF, GLS, parameters of diastolic function)
* Thrombotic complications, cardiovascular events, hospitalizations

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Documented SARS-COV-2 infection with PCR test
* Need for hospitalization in a COVID clinic
* Informed written consent

Exclusion Criteria:

* Inability to cooperate for peripheral arterial tonometry
* Hemodynamic instability
* High probability of non-compliance with the procedures of the study
* Reduced life expectancy <1 year
* Established atherosclerotic cardiovascular disease
* Pregnancy, postpartum
* Alcoholism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients who developed COVID-19 disease for which admission for hospitalization was required, while the control group will be healthy matched volunteers for age, gender and cardiovascular risk factors.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Natural logarithm of reactive hyperemia index (Ln-RHI) | 2 months after discharge
  Endothelial dysfunction is defined as LnRHI≤0.51

SECONDARY OUTCOMES:
Area under the Curve (AUC) of the Reactive Hyperemia index (RHI) measurements during hospitalization, at 2 months after discharge and at 6 months after discharge. | At 6 months after discharge
Natural logarithm of reactive hyperemia index (Ln-RHI) | During hospitalization (up to day 10)
Reactive Hyperemia Index (RHI) | At 6 months after discharge
Rate of endothelial dysfunction (LnRHI≤0.51) | During hospitalization (up to day 10)
Rate of endothelial dysfunction (LnRHI≤0.51) | At 2 months after discharge
Rate of endothelial dysfunction (LnRHI≤0.51) | At 6 months after discharge
Change in RHI index (ΔRHI) from hospitalization to 6 months | At 6 months after discharge
Duration (days) of hospitalization for COVID-19 | Predischarge (up to 3 months)
Incidence of thrombotic events | Up to 12 months after discharge
Incidence of cardiovascular events | Up to 12 months after discharge
Mortality | Up to 12 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Moulias, MD, PhD, Principal Investigator — General University Hospital of Patras; Periklis Davlouros, MD, PhD, Principal Investigator — General University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No